CLINICAL TRIAL: NCT03760445
Title: A Phase I/II Multi-center Study of HDM201 Added to Chemotherapy in Adult Subjects With Relapsed/Refractory (R/R) or Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: HDM201 Added to CT in R/R or Newly Diagnosed AML
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: It was determined that the study design may not be optimal given the changing AML treatment landscape.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHDM201A2101; 2018-003107-19 (EudraCT Number)
Record Dates: First submitted 2018-11-13; First posted 2018-11-30 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: HDM201; midostaurin; cytarabine; daunorubicin; idarubicin; liposomal cytarabine/daunorubicin; acute myeloid leukemia (AML); 1L newly diagnosed AML; relapsed/refractory AML; FLT3-mutation; combination treatment; dose escalation; CR/CRi; minimal residual disease; DDI with CYP3A4 inhibitors; DDI with sensitive CYP3A4 substrate
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — siremadlin; Cytarabine; Anthracyclines; Daunorubicin; Idarubicin; midostaurin; posaconazole; Midazolam

STUDY DESIGN:
Intervention Model Description: 3 parts - two different populations Part 1 - escalation - parallel dose escalation in 1L AML subjects and in R/R subjects (up to 8 dose cohorts per arm.
  Part 2 - expansion - parallel expansion in 3 cohorts of 1L AML, and 1 cohort of R/R AML after recommended dose of expansion was determined.
  Part 3 - DDI - parallel enrollment or R/R AML subjects into 2 DDI Cohorts (one with CYP3A4 inhibitor, one with CYP3A4 substrate).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1 - first line (1L) AML (Experimental): 1L acute myeloid leukemia (AML) subjects receiving HDM201 in various doses/schedules in combination with cytarabine/anthracyclines
  Interventions: Drug: HDM201; Drug: cytarabine; Drug: anthracycline
- Part 1 - relapsed/refractory (R/R) AML (Experimental): R/R AML subjects receiving HDM201 in various doses/schedules in combination with cytarabine
  Interventions: Drug: HDM201; Drug: cytarabine
- Part 2 - Expansion Cohort 1 (Experimental): 1L de novo AML subjects without documented FLT3 mutation receiving HDM201 at the recommended dose of expansion (RDE) in combination with cytarabine/anthracyclines
  Interventions: Drug: HDM201; Drug: cytarabine; Drug: anthracycline
- Part 2 - Expansion Cohort 2 (Experimental): 1L de novo AML subjects with documented FLT3 mutation status receiving HDM201 at RDE in combination with cytarabine/anthracyclines and midostaurin
  Interventions: Drug: HDM201; Drug: cytarabine; Drug: anthracycline; Drug: midostaurin
- Part 2 - Expansion Cohort 3 (Experimental): 1L secondary AML subjects receiving HDM201 at RDE in combination with liposomal cytarabine/daunorubicin
  Interventions: Drug: HDM201; Drug: cytarabine; Drug: liposomal cytarabine/daunorubicin
- Part 2 - Expansion Cohort 4 (Experimental): R/R AML subjects receiving HDM201 at RDE in combination with cytarabine
  Interventions: Drug: HDM201; Drug: cytarabine
- Part 3 - DDI Cohort 1 (Experimental): R/R AML subjects receiving HDM201 at adjusted recommended Phase 3 dose (RP3D) determined in Part 2 in combination with cytarabine and posaconazole added in Cycle 1
  Interventions: Drug: HDM201; Drug: cytarabine; Drug: posaconazole
- Part 3 - DDI Cohort 2 (Experimental): R/R AML subjects receiving HDM201 at RP3D in combination with cytarabine and midazolam
  Interventions: Drug: HDM201; Drug: cytarabine; Drug: midazolam

INTERVENTIONS:
Drug: HDM201 — 2.5 mg and 10mg capsules, given orally
  Other Names: none available
Drug: cytarabine — 20mg or 1000 mg or other strengths as locally available given intravenously
  Other Names: Ara-C, Cytosar
Drug: anthracycline — 20mg or other strength as locally available given intravenously
  Other Names: daunorubicin or idarubicin, Rubidomycin or Idamycin
  Arms: Part 1 - first line (1L) AML; Part 2 - Expansion Cohort 1; Part 2 - Expansion Cohort 2
Drug: midostaurin — 25mg capsules given orally
  Other Names: PKC412, Rydapt
  Arms: Part 2 - Expansion Cohort 2
Drug: liposomal cytarabine/daunorubicin — 100mg/44mg or other strength as locally available given intravenously
  Other Names: Vyxeos
  Arms: Part 2 - Expansion Cohort 3
Drug: posaconazole — 100mg delayed release tablet or other strength as locally available given orally
  Other Names: Noxafil
  Arms: Part 3 - DDI Cohort 1
Drug: midazolam — 2mg/mL oral solution or in other strength as locally available
  Other Names: midazolam HCl
  Arms: Part 3 - DDI Cohort 2

SUMMARY:
This is a multi-center open-label Phase I/II study investigating orally administered HDM201 in combination with chemotherapy in two populations: subjects with first line AML or subjects with relapsed/refractory AML. This study is conducted in three parts: dose escalation, dose expansion and DDI study.

DETAILED DESCRIPTION:
This is a Phase 1 / 2 study. No patients were screened / enrolled. There are no data collected. There will be no CSR.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Signed informed consent must be obtained prior to participation in the study
* Age ≥18
* Diagnosis of AML based on WHO 2016 classification. Patients with APL (acute promyelocytic leukemia) with PML-RARA are not eligible.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) that is 0 - 2.
* Adequate organ functions
* Left ventricular ejection fraction > 45%

For 1L AML population:

* For Part 1 or Part 2 Expansion Cohorts 1 or 2: subjects with de novo AML suitable for induction treatment with cytarabine and anthracyclines as per investigator judgement
* For Part 2 Expansion Cohort 2: documented presence of FLT3 mutation (ITD or TKD ) and suitable for midostaurin treatment as per investigator judgement.
* For Part 2 Expansion Cohort 3: Subjects with secondary AML (e.g. AML-MRC , secondary to myelodysplasia/MDS or therapy-related AML). Prior use of hypomethylating agents or other therapies with curative intent for treatment previous hematological malignancies or therapy-related AML is allowed. Subjects suitable for induction treatment with liposomal cytarabine/daunorubicin as per investigator judgement.

For R/R AML population:

* All Parts: Diagnosis of relapsed or refractory AML and suitable for treatment with IDAC as per investigator judgement.
* For Part 3 only: willingness and suitability to participate in DDI Cohort 1 or 2.

Exclusion Criteria:

* Prior exposure to MDM2 and MDM4 inhibitor (e.g. idasanutlin)
* Known symptomatic CNS leukemia not controlled by adequate therapy.
* Isolated extramedullary leukemia
* Subjects with prior malignancy (some exceptions apply)
* QTcF > 470 ms at screening
* Subjects who require treatment with moderate or strong CYP3A4 inducers within 14 days prior to starting study treatment or during the study
* Subjects who require use of herbal preparations/medications and dietary supplements within 7 days prior to first dose and during the study
* Subjects who require treatment with substrates of CYP3A4/5 with narrow therapeutic index (within 24 hours prior to during and 48 hours after HDM201 administration)
* Subjects who require treatment with moderate or strong CYP3A4 inhibitors within 48 hours prior to, during and 48 hours post HDM201 administration. (except for Part 3 DDI Cohort 1 and 2)
* Subject is pregnant or breastfeeding
* WOCBP unless using highly effective methods of contraception during study treatment and for an appropriate time period after last study treatment
* Sexually active males unless they use a condom during intercourse while taking study drug and for an appropriate time period after last study treatment

For Part 1 only:

- Subjects with a known favorable risk AML subtype at screening or subjects with FLT3 mutation

For Part 3 only:

* DDI Cohort 1: use of posaconazole (other than the planned dosing required by the protocol) within 7 days prior to start of the DDI investigation and for the duration of the DDI period
* DDI Cohort 2: use of midazolam (other than the planned dosing required by the protocol) within 2 days prior to start of the DDI investigation and for the duration of the DDI period
* DDI Cohort 1 and 2: subjects who have received, or are expected to receive moderate or strong inhibitors of CYP3A4 within 7 days prior to start of the DDI investigation, for the duration of the investigation, and 24 hours after last blood sample collection for PK assessment

Other protocol-defined inclusion/exclusion may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2021-07-22 (Estimated); Study Completion 2023-06-13 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Incidence of dose limiting toxicity (DLT) | first day of study treatment to 3 months after start of study treatment
  number of DLTs by dose regimen of first line (1L) acute myeloid leukemia (AML) subjects during induction treatment; number of DLTs by dose regimen of relapsed/refractory (R/R) AML subjects during treatment
Part 1 - Time to DLT | first day of study treatment to 3 months after start of study treatment
  time from first dose to onset of DLT by dose regimen of 1L AML and R/R AML subjects
Part 1 - Incidence and severity of Adverse Events (AEs) | first day of study treatment to 3 months after start of study treatment
  number and grade of AEs by dose regimen of 1L AML and R/R AML subjects during DLT observation period
Part 2 - Incidence and severity of AEs/serious adverse events (SAEs) | first day of study treatment until 8.5 months after start of study treatment
  number and grade of AEs/SAEs by expansion cohort
Part 2 - Percentage of participants with complete remission (CR)/CR with incomplete recovery (CRi) with adequate blood count recovery (ABCR) | first day of study treatment until 4.5 months after start of study treatment
  Percentage of participants with CR/CRi with ABCR at the end of induction treatment for Expansion Cohort 1, and at the end of treatment for Expansion Cohort 4
Part 2 - Incidence and severity of abnormal laboratory values | first day of study treatment until 8.5 months after start of study treatment
  number and grade of abnormal laboratory results by expansion cohort
Part 2 - Incidence and severity of abnormal electrocardiogram (ECG) results | first day of study treatment until 8.5 months after start of study treatment
  number and severity of abnormal ECG results by expansion cohort
Part 2 - Incidence and severity of abnormal vital signs | first day of study treatment until 8.5 months after start of study treatment
  number and severity of abnormal vital signs by expansion cohort
Part 3 - DDI Cohort 1 HDM201 Pharmacokinetics (PK) area under the curve (AUC) | first day of HDM201 dose to 10 days after start of HDM201
  determine HDM201 AUC from time zero to the last measurable concentration sampling time (AUClast) in Cycle 1
Part 3 - DDI Cohort 1 HDM201 PK maximum observed plasma concentration (Cmax) | first day of HDM201 dose to 10 days after start of HDM201
  determine HDM201 Cmax in Cycle 1
Part 3 - DDI Cohort 1 HDM201 PK average plasma concentration | first day of HDM201 dose to 10 days after start of HDM201
  determine HDM201 average plasma concentration in Cycle 1
Part 3 - DDI Cohort 1 HDM201 PK time of maximum observed plasma concentration (Tmax) | first day of HDM201 dose to 10 days after start of HDM201
  determine HDM201 Tmax in Cycle 1
Part 3 - DDI Cohort 2: midazolam PK AUC | first dose of midazolam (Day-2) to 8 days after start of study treatment (HDM201)
  determine midazolam AUC last and AUC from time zero to infinity (inf)
Part 3 - DDI Cohort 2: midazolam PK Cmax | first dose of midazolam (Day-2) to 8 days after start of study treatment (HDM201)
  determine midazolam Cmax

SECONDARY OUTCOMES:
Part 1 +2: HDM201 PK AUC | first day of study treatment to 7.5 months after start of study treatment
  determine HDM201 AUC by dose regimen in Part 1, and Expansion Cohort in Part 2
Part 1 +2: HDM201 PK Cmax | first day of study treatment to 7.5 months after start of study treatment
  determine Cmax of HDM201 by dose regimen in Part 2, and Expansion Cohort in Part 2
Part 1 +2: HDM201 PK Tmax | first day of study treatment to 7.5 months after start of study treatment
  determine Tmax of HDM201 by dose regimen in Part 2, and Expansion Cohort in Part 2
Part 1 - incidence of AEs/SAEs | first day of study treatment to 8.5 months after start of study treatment
  number and grade of AEs/SAEs, by dose regimen for 1L AML and R/R AML subjects during study treatment + 30 days
Part 2 - all Expansion Cohorts: time to platelet recovery | first day of study treatment to 7.5 months after start of study treatment
  determine time to platelet recovery by Expansion Cohort for each cycle
Part 2 - all Expansion Cohorts: time to neutrophil recovery | first day of study treatment to 7.5 months after start of study treatment
  determine time to neutrophil recovery by Expansion Cohort for each cycle
Part 2 - all Expansion Cohorts: overall survival | first day of study treatment to 3 years after last patient is enrolled to Part 2
  determine overall survival by Expansion Cohort
Part 2 - all Expansion Cohorts: event-free survival | first day of study treatment to 3 years after last patient is enrolled to Part 2
  determine event-free survival by Expansion Cohort
Part 2 - all Expansion Cohorts: Percentage of subjects receiving Hematopoietic stem cell transplant (HSCT) | first day of study treatment to 3 years after last patient was enrolled to Part 2
  percentage of subjects receiving HSCT after study treatment by Expansion Cohort.
Part 2 - Expansion Cohorts 1 to 3: disease-free survival (DFS) | first day of study treatment to 3 years after last patient enrolled to Part 2
  determine DFS by Expansion Cohort
Part 2 - Expansion Cohorts 1 to 3: cumulative incidence of relapse (CIR) | first day of study treatment to 3 years after last patient enrolled to Part 2
  determine CIR by Expansion Cohort
Part 2 - Expansion Cohorts 2 and 3 - proportion of subjects with CR/CRi with ABCR | first day of study treatment to 7.5 months after start of study treatment
  proportion of subjects achieving CR or CRi with ABCR by Expansion Cohort
Part 2 - Expansion Cohorts 1 and 2: proportion of subjects with minimal/measurable residual disease (MRD) negativity | first day of study treatment to 7.5 months after start of study treatment
  proportion of subjects achieving MRD negativity by Expansion Cohort
Part 2 - expansion cohort 2: midostaurin PK AUC | first day of study treatment to 7.5 month after start of study treatment
  determine midostaurin AUC
Part 2 - expansion cohort 2: midostaurin PK Cmax | first day of study treatment to 7.5 month after start of study treatment
  determine midostaurin Cmax during induction and consolidation treatment
Part 2 - expansion cohort 2: midostaurin PK Tmax | first day of study treatment to 7.5 month after start of study treatment
  determine midostaurin Tmax during induction and consolidation treatment
Part 1 - incidence of abnormal laboratory values | first day of study treatment to 8.5 months after start of study treatment
  number of abnormal laboratory results by dose regimen for 1L AML and R/R AML subjects during study treatment + 30 days
Part 1 - incidence of abnormal ECG results | first day of study treatment to 8.5 months after start of study treatment
  number of abnormal ECG results by dose regimen for 1L AML and R/R AML subjects during study treatment + 30 days
Part 1 - incidence of abnormal vital signs | first day of study treatment to 8.5 months after start of study treatment
  number of abnormal vital signs by dose regimen for 1L AML and R/R AML subjects during study treatment + 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.